CLINICAL TRIAL: NCT02910427
Title: The Effect of Intervention With Potassium and/ or Magnesium-enriched Salt on Neurological Performance of Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academia Sinica, Taiwan (Other)
Responsible Party: Principal Investigator, Wen-Harn Pan, Research Fellow, Academia Sinica, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AS-IRB-BM-08013
Record Dates: First submitted 2016-09-09; First posted 2016-09-22 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-09

CONDITIONS: Stroke
Keywords: stroke; potassium and magnesium-enriched salt; neurological performance
MeSH Terms: conditions — Stroke | interventions — Potassium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Na salt (Placebo Comparator): regular salt
  Interventions: Other: Regular salt
- K salt (Active Comparator): potassium-enriched salt
  Interventions: Other: Potassium-enriched salt
- K/Mg salt (Active Comparator): potassium and magnesium-enriched salt
  Interventions: Other: Potassium and magnesium-enriched salt

INTERVENTIONS:
Other: Regular salt — Participants eat a regular salt diet.
  Arms: Na salt
Other: Potassium-enriched salt — Participants eat a potassium-enriched salt diet.
  Arms: K salt
Other: Potassium and magnesium-enriched salt — Participants eat a potassium and magnesium-enriched salt diet.
  Arms: K/Mg salt

SUMMARY:
Cerebrovascular disease is the second leading cause of death in Taiwan. Although stroke incidence and mortality decline steadily in Taiwan, its impact on medical cost, quality of life and neurological deficits remains extraordinary. Stroke incidence and mortality are also rising in the developed countries presumably due to a world-wide increase in prevalence of obesity and metabolic syndrome. Negative associations have been observed between high blood pressure, hyperglycemia and two major dietary cations in vegetables and dairy products: potassium and magnesium. Mean levels of dietary potassium and magnesium intake in Taiwan are much lower than those of dietary reference intake. Short term supplementation studies have demonstrated their effects in reducing blood pressure and degree of insulin resistance. However, long-term studies on cardiovascular events are lacking. Our previous long-term intervention trial in elderly veteran home showed a 41% reduction in cardiovascular mortality by simply switching regular cooking salt to potassium-enriched salt in kitchens. The investigators have previously observed an annual reduction of medical cost around $ 15,000 NT in the aforementioned veteran home trial. A multi-centered randomized controlled trial was carried out with three arms: (1) regular salt (Na salt), (2) potassium-enriched salt (K salt), and (3) potassium and magnesium-enriched salt (K/Mg salt). The objectives of this study was to investigate whether potassium and magnesium-enriched salt would improve the neurological performance of the stroke patients.The investigators anticipate to observe beneficial effect from consuming potassium and magnesium enriched salt for neurological improvement in stroke patients.

ELIGIBILITY:
Inclusion Criteria:

1. hospitalization within 1 month due to cerebral infarction or hemorrhage;
2. a modified Rankin Score of 4 or less at the time of discharge;
3. an age of 45 or older; and
4. an agreement to prepare foods with salt provided by the project.

Exclusion Criteria:

1. patients with poor kidney function (glomerular filtration rate<60 ml/min), secondary hypertension, cancer, or liver diseases;
2. patients with eating disorders;
3. patients taking K-sparing medicines;
4. or patients using salt substitutes.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 291 (Actual)
Dates: Start 2009-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
The modified Rankin scale (mRs) | 6 months
The National Institute of Health Stroke Scale (NIHSS) | 6 months
The Barthel index (BI) | 6 months
The "good neurological performance" | 6 months
  The "good neurological performance" is defined as those who met all of the following criteria: a score of zero in NIHSS, a score of 100 in BI, and a score of equal to or less than 1 in mRS.

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Harn Pan, Ph.D., Principal Investigator — Institute of Biomedical Sciences, Academia Sinica

REFERENCES:
- [Derived] Pan WH, Lai YH, Yeh WT, Chen JR, Jeng JS, Bai CH, Lin RT, Lee TH, Chang KC, Lin HJ, Hsiao CF, Chern CM, Lien LM, Liu CH, Chen WH, Chang A. Intake of potassium- and magnesium-enriched salt improves functional outcome after stroke: a randomized, multicenter, double-blind controlled trial. Am J Clin Nutr. 2017 Nov;106(5):1267-1273. doi: 10.3945/ajcn.116.148536. Epub 2017 Sep 6. PMID 28877896